CLINICAL TRIAL: NCT07175558
Title: Effects of Reiki Applied to Patients Undergoing Colorectal Cancer Surgery on Postoperative Pain, Anxiety, Physiological Parameters and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sena Melike Tasci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RPAPR
Record Dates: First submitted 2024-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Reiki; Nursing care; Surgical Nursing; Colorectal Cancer Surgery; Physiological Parameters
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial with an intervention and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reiki Group (Experimental): The patient will be explained about reiki (life energy recovery) and the application environment will be kept quiet. Metal objects on the patient and the researcher will be removed. The researcher will wash and warm their hands. The patient's privacy will be ensured. The patient will be given a flat lying position with their arms and legs on both sides and comfortable. The patient will be asked to close their eyes. The researcher's fingers will be straight, side by side and closed, and energy will be provided to the application areas; crown chakra (top of the head), forehead chakra (top of the forehead), throat chakra (top of the throat), heart chakra (middle of the chest), solar plexus (under the chest, above the navel), sacral chakra (below the navel) and root chakra (upper back). Reiki application will be applied to the points on the 7 chakra regions for 4 minutes each, for a total of 28 minutes. The patient will be asked to open their eyes at the end of the application.
  Interventions: Other: Reiki
- Control Group (No Intervention): The control group will not receive any intervention and will receive care in accordance with the clinic's own schedule.

INTERVENTIONS:
Other: Reiki — The patient will be explained about reiki (life energy recovery) and the application environment will be kept quiet.
  Metal objects on the patient and the researcher will be removed. The researcher will wash and warm their hands. The patient's privacy will be ensured. The patient will be given a flat lying position with their arms and legs on both sides and comfortable. The patient will be asked to close their eyes. The researcher's fingers will be straight, side by side and closed, and energy will be provided to the application areas; crown chakra (top of the head), forehead chakra (top of the forehead), throat chakra (top of the throat), heart chakra (middle of the chest), solar plexus (under the chest, above the navel), sacral chakra (below the navel) and root chakra (upper back). Reiki application will be applied to the points on the 7 chakra regions for 4 minutes each, for a total of 28 minutes. The patient will be asked to open their eyes at the end of the application.
  Arms: Reiki Group

SUMMARY:
Reiki touch therapy has been used for many years, especially on pain, anxiety and physiological parameters, and studies have been found to show that it is effective. In a systematic review conducted with Sectio patients, it was determined that reiki reduces pain. In a study conducted by Zare et al. with patients undergoing coronary bypass surgery, it was reported that reiki regulates the respiratory rate. It was determined that reiki applied to the incision area in patients undergoing abdominal surgery reduces pain. In a different study, it was emphasized that reiki applied to 90 women who gave birth by cesarean section in the experimental group on the 1st and 2nd days after surgery decreased pain and anxiety levels, analgesic requirement and respiratory rate after surgery compared to the control group, while there was no change in blood pressure and pulse. In a meta-analysis study including four studies consisting of 104 patients in the Reiki group and 108 patients in the control group, a statistically significant decrease in the pain score of the Reiki group was found. In a study conducted by Bremner and colleagues, it was determined that stress, anxiety and depression decreased in the Reiki group. In a study measuring the effect of Reiki use on pain, stress and anxiety levels in patients undergoing total knee replacement surgery, significant decreases were found in pain, blood pressure, respiratory rate and anxiety levels in the Reiki group out of three groups that received Reiki, sham Reiki and standard care. In line with these studies, evidence-based data on the effectiveness of Reiki is thought to help nurses reduce patients' postoperative pain and anxiety, reduce the incidence of respiratory complications and help them evaluate and manage physiological parameters more accurately.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteer to participate and continue in the study,
* Have no communication problems that would prevent the interview,
* Have pain levels of 5 and above according to the GKO,
* Have no history of psychiatric disorders and therefore do not use medication will be included in the study.

Exclusion Criteria:

* If a different surgical procedure is performed other than colorectal surgery,
* If the score determined in the Visual Comparison Scale in the pre-operative evaluation of the patient is 7 and above,
* If there is cancer pain,
* If there are complex cancer metastases,
* If there are secondary metastases from colorectal cancer,
* If there is persistent severe nausea and vomiting during the procedure and post-operative period,
* If the patient is illiterate,
* If the patient is over 50 points from the Trait Anxiety Scale,
* If the patient has had abdominal surgery before,
* If the patient has had reiki or energy therapies before,
* If the patient is using medications other than the routine treatment after the surgery, the patients will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Pain NRS Scale: Time 1 | Before surgery
  The pain experienced should be numbered on a linear line and rated as "none, mild, moderate, or severe." A rating of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain.
Pain NRS Scale: Time 2 | 4th hour after surgery
  The pain experienced should be numbered on a linear line and rated as "none, mild, moderate, or severe." A rating of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain.
Pain NRS Scale: Time 3 | 1st day after surgery
  The pain experienced should be numbered on a linear line and rated as "none, mild, moderate, or severe." A rating of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain.
Pain NRS Scale: Time 4 | 2nd day after surgery
  The pain experienced should be numbered on a linear line and rated as "none, mild, moderate, or severe." A rating of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain.
State-Trait Anxiety Inventory: Time 1 | Before surgery
  Developed by Spielberger, Gorsuch, and Lushene in 1970, the scale consists of two subscales with 20 items each measuring state and trait anxiety. The STAI used in this study is answered using a 4-point Likert scale. The emotions and behaviors expressed in the STAI items are indicated by selecting one of the following options: (1) Not at all, (2) A little, (3) A lot, and (4) Completely, according to the severity of such experiences. High scores on the scale indicate high levels of anxiety The highest score is 80, and the lowest is 20. The higher the total anxiety score, the higher the person's anxiety level is interpreted. . The adaptation, validity, and reliability study of the scale was conducted into Turkish by Öner and Le Compte in 1983. Cronbach's α internal consistency rate for the scale's current sample was found to be 0.90 for the State Anxiety Scale.
State-Trait Anxiety Inventory: Time 2 | 2nd day after surgery
  Developed by Spielberger, Gorsuch, and Lushene in 1970, the scale consists of two subscales with 20 items each measuring state and trait anxiety. The STAI used in this study is answered using a 4-point Likert scale. The emotions and behaviors expressed in the STAI items are indicated by selecting one of the following options: (1) Not at all, (2) A little, (3) A lot, and (4) Completely, according to the severity of such experiences. High scores on the scale indicate high levels of anxiety The highest score is 80, and the lowest is 20. The higher the total anxiety score, the higher the person's anxiety level is interpreted. The adaptation, validity, and reliability study of the scale was conducted into Turkish by Öner and Le Compte in 1983. Cronbach's α internal consistency rate for the scale's current sample was found to be 0.90 for the State Anxiety Scale.
Postoperative Recovery Index | 15th day after surgery
  The postoperative recovery index, the validity and reliability of which was conducted by Butler et al. (2012), consists of 25 items. The ASII has five subdimensions: psychological symptoms, physical activities, general symptoms, bowel symptoms, and desire symptoms. In scoring the questionnaire, the scores of the items in the subdimensions are summed, their arithmetic means are taken, and the subdimension score is determined. To obtain the total score of the ASII survey, all 25 items are summed and their arithmetic mean is taken. High scores on the index reflect more difficulties in postoperative recovery, while low scores indicate that postoperative recovery was easier. In this study, the ASII, the validity and reliability of which was conducted for Turkish by Hande Cengiz in 2018, was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Eğitim ve Araştırma Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study can be shared after completion if requested by the reader.

REFERENCES:
- [Background] 1. Thrane, S, Cohen, SM. Effect of Reiki therapy on pain and anxiety in adults: an in-depth literature review of randomized trials with effect size calculations. Pain management nursing, 2014,15(4), 897-908. 2. Zare, Z. Shahsavari, H, Moeini, M. Effects of therapeutic touch on the vital signs of patients before coronary artery bypass graft surgery. Iranian Journal of Nursing and Midwifery Research. 2010;15(1), 37-42. 3. 3. Sagkal Midilli, T. Ciray Gunduzoglu, N. Effects of reiki on pain and vital signs when applied to the ıncision area of the body after cesarean section surgery: A single-blinded, randomized, double-controlled study. Holistic Nursing Practice. 2016;30(6), 368-378. 4. Demirdogan M. The effect of Reiki on pain: A meta-analysis. Complementary Therapies in Clinical Practice. 2018;31, 384-387 5. Baldwin AL, Vitale A, Brownell E, Kryak E, Rand W. Effects of reiki on pain, anxiety, and blood pressure in patients undergoing kneere placement. Holistic Nursing Practice. 2017;31(2): 80-89. 6. Keşer, E, Bağlama, SS, Sezer, C. The effect of reiki and aromatherapy on vital signs, oxygen saturation, and anxiety level in patients undergoing upper gastrointestinal endoscopy: A randomized controlled study. Holistic Nursing Practice, 2023;37(6):337-346. 7. Şişman, H, Arslan, S. The effect of reiki on anxiety, fear, pain, and oxygen saturation in abdominal surgery patients: A randomized controlled trial. Explore. 2023;19(4), 578-586. 8. Yeşil Bayülgen, M, Gün, M. The effect of Reiki on fatigue and comfort in hemodialysis patients. Explore. 2023;19(4):553-560.